CLINICAL TRIAL: NCT04767932
Title: Investigation of Impacts of Vibration on Muscular Strength and Functional Performance of Upper Limbs of Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N201907023
Record Dates: First submitted 2020-11-12; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control group (Experimental): the control group will receive regular exercise training at same time.
  Interventions: Behavioral: vibration machine

INTERVENTIONS:
Behavioral: vibration machine — Experimental: vibration intervention the experimental group will perform 20mins/ section, three times weekly for 8 weeks vibration training

SUMMARY:
The elderly population is increasing at worldwide. The need of health promotion and maintenance for elderly adults has become a critical issue. According to a national investigation in 2017, the number of people over 65 years old accounts for 13.33% of the total population and would reach 20.1% by 2050. Muscle strength and functional performances of upper limbs play an important role in most daily activities in elderly adults. However, with aging, the muscle strength of upper extremities could be affected and decrease the functional performances of daily living. Vibration exercise can be used to induce the muscle contraction and motor control in lower limbs for people with neuromuscular disorders. Few studies have investigated the training effects on muscle strength and functional performances of upper limbs for elderly adults。Therefore, appropriate training devices and exercise programs to facilitate the muscle strength and functional performances of upper limbs in elderly people would be needed for clinical therapists. Therefore, the purpose of this study was to develop a vibration training device and investigate the training effects on muscle strength and functional performances of upper limbs in elderly people. This study will recruit 44 elderly adults, evaluating the muscle strength and functional performances of upper limbs before and after interventions. All subjects will be randomized assign to experimental and control groups; the experimental group will perform 30mins/ section, three times weekly for 8 weeks vibration training, and the control group will receive regular exercise training at same time. Two-way ANOVA with repeated measure will be applied to analyze the training effects and difference in the muscle strength and functional performances of upper limbs between two groups. SPSS version 18.0 statistical software will be used. The α level for statistical significance is set at 0.05.

DETAILED DESCRIPTION:
Vibration exercise can be used to induce the muscle contraction and motor control in lower limbs for people with neuromuscular disorders. Few studies have investigated the training effects on muscle strength and functional performances of upper limbs for elderly adults。Therefore, appropriate training devices and exercise programs to facilitate the muscle strength and functional performances of upper limbs in elderly people would be needed for clinical therapists. Therefore, the purpose of this study was to develop a vibration training device and investigate the training effects on muscle strength and functional performances of upper limbs in elderly people. This study will recruit 44 elderly adults, evaluating the muscle strength and functional performances of upper limbs before and after interventions. All subjects will be randomized assign to experimental and control groups; the experimental group will perform 30mins/ section, three times weekly for 8 weeks vibration training, and the control group will receive regular exercise training at same time. Two-way ANOVA with repeated measure will be applied to analyze the training effects and difference in the muscle strength and functional performances of upper limbs between two groups. SPSS version 18.0 statistical software will be used. The α level for statistical significance is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

Sarcopenia of older people

Exclusion Criteria:

1. Upper limbs acute or chronic nerve, musculoskeletal injury within 6 months
2. Upper extremity surgery in 6 months
3. without a pacemaker
4. without severe vision or hearing problems
5. without severe heart disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
muscle strength of upper limbs. | 15 min
  use MicroFET3 to understand physical fitness of upper limbs between groups after intervention .The tool for assessing upper limb muscle strength is a tool with good reliability and validity. It includes wrist flexor, extensor, brachioradialis, biceps, triceps, and deltoid muscle strength performance. The researcher places the muscle to be measured and asks the subject to hold the dynamometer for three to five seconds, measure twice, record in kilograms to one decimal place, and measure twice in total. The higher value is recorded in kilograms to the next decimal place.

SECONDARY OUTCOMES:
Assess the improvement of quality of life due to muscle strength improvement | 20 min
  IADL+ Quality of life to understand physical fitness and functional performance of upper limbs between groups after intervention .This sub-questionnaire is based on the subjective feelings of the elderly in the last two weeks, measured by interviews and observation behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: chia-hui kao, master, Principal Investigator — student
Locations (1):
- TMU, Taipei, Taiwan